CLINICAL TRIAL: NCT03472690
Title: A Phase 2, Multi-center, Randomized, Double-Blind, Placebo-Controlled Study of QBECO SSI for the Induction and Maintenance of Clinical and Endoscopic Remission in Subjects With Moderate to Severe Crohn's Disease
Brief Title: QBECO SSI for Clinical and Endoscopic Remission in Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate Decision to terminate study after Lead-In portion of the study completed.
Sponsor: Qu Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QBECO-CD-02
Record Dates: First submitted 2018-03-08; First posted 2018-03-21 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Disease 1
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage one is Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): 0.1 mL, self-administered subcutaneous injection, every second day
  Interventions: Biological: QBECO-SSI
- Placebo (Placebo Comparator): 0.1 mL, self-administered subcutaneous injection, every second day
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: QBECO-SSI — Subcutaneous injection
  Arms: Active
Other: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The QBECO-CD-02 trial in subjects with moderate to severe Crohn's disease (CD) is intended to build on past experience with QBECO SSI and further establish the safety and efficacy of QBECO SSI for the induction of clinical and/or endoscopic response and remission.

The study will be conducted in three stages; a Lead-in, Main Induction and Main Maintenance .The first 20 patients will be enrolled in the Lead-in study, at approximately 5 study centers in Canada. Subsequent patients will be enrolled in the Main study, which aims to enroll 150 patients. The Lead-in component will be an open-label study to evaluate endoscopic healing endpoints. The Main Induction study will be randomized and placebo-controlled. Participants meeting response criteria following the Main Induction study will be eligible to continue into the Main Maintenance study, remaining on their initially randomized treatment. Participants not meeting response criteria will complete their follow-up and study involvement at the end of the Main Induction.

DETAILED DESCRIPTION:
The QBECO-CD-02 trial in subjects with moderate to severe Crohn's disease (CD) is intended to build on past experience with QBECO SSI and further establish the safety and efficacy of QBECO SSI for the induction of clinical and/or endoscopic response and remission.

i. Overall Design:

Phase II, randomized, double-blind, placebo-controlled study in subjects with moderate to severe Crohn's disease to establish the safety and efficacy of QBECO SSI for the induction and maintenance of clinical and/or endoscopic response and remission. The study will be conducted in three stages; a Lead-in, Main Induction and Main Maintenance . The first 20 patients will be enrolled in the Lead-in study, at selected study centers. Subsequent patients will be enrolled in the Main study. The Lead-in component will be an open-label study to evaluate endoscopic healing endpoints. The Main Induction study will be randomized and placebo-controlled. Participants meeting response criteria following the Main Induction study will be eligible to continue into the Main Maintenance study, remaining on their initially randomized treatment. Participants not meeting response criteria will complete their follow-up and study involvement at the end of the Main Induction.

Primary Endpoints will be evaluated at various times throughout each stage of the study. In the Lead-In study, primary endpoints will be measured at Week 16 and 26 for determination of the induction duration and again at Week 52 as initial data on maintenance. In the Main Induction, the primary endpoints will be assessed when the last subject completes the induction period, either Week 16 or Week 26 depending on the finding of the Lead-In. In the Main Maintenance, the primary endpoints will be measured at Week 52. Safety Assessments will be carried out throughout the study and at the Week 56 visits for all subjects completing the study.

The study will be run at approximately 50 study centers in Canada, the United States of America and Eastern Europe.

ii. Number of Participants:

20 participants will be enrolled in the Lead-In study. No Lead-In study participants will be enrolled in the Main Induction or Maintenance component of the study.

150 participants will be randomized to the Main Induction study, resulting in an estimated total of 70 subjects proceeding to the Main Maintenance component of the study.

iii. Intervention Groups and Duration:

Approximately 170 adult subjects (N=170) with moderate to severe CD, 20 patients in the Lead-In study and 150 patients in the Main study, stratified by prior anti-TNFα inhibitor/ biologic therapy use. Patients will be randomized 2:1, active drug:placebo, and will receive 52 weeks of QBECO SSI treatment or placebo.

iv. Objectives and Endpoints:

Lead-In:

1. Primary

   1. To determine whether Week 26 provides superior endoscopic healing outcomes compared to Week 16
   2. To evaluate the incidence of adverse events (safety & tolerability) as measured by frequency and severity of adverse events.
2. Secondary

   1. To determine the effect of QBECO SSI on endoscopic remission at the end of 52 weeks of treatment
   2. To determine the effect of QBECO SSI on clinical remission, as measured by abdominal pain and soft-stool frequency, at the end of the induction period

Main:

* Induction:

  1. Primary

     1. To determine the effect of QBECO SSI on clinical remission, as measured by abdominal pain and soft-stool frequency, at the end of the induction period
     2. To determine the effect of QBECO SSI on endoscopic remission at the end of the induction period
     3. To evaluate the incidence of adverse events (safety and tolerability) as measured by frequency and severity of adverse events.
  2. Secondary

     1. To determine the effect of QBECO SSI on abdominal pain score at the end of the induction period (i.e., change from baseline)
     2. To determine the effect of QBECO SSI on soft-stool score at the end of the induction period (i.e., change from baseline)
     3. To determine the effect of QBECO SSI on endoscopic response at the end of the induction period
     4. To determine the effect of QBECO SSI on Simple Endoscopic Score for Crohn's Disease (SES-CD) scores at the end of the induction period as defined by SES-CD reduction by ≥25% and ≥75% and change from baseline
     5. To determine the effect of QBECO SSI on histological activity at the end of induction period as defined by 25%, 50% and 75% reduction in global colonic Global Histologic Disease Activity Score (GHAS) and Robarts Histological Index (RHI)
     6. To determine the effect of QBECO SSI on simultaneous clinical and endoscopic remission at the end of the induction period
* Maintenance:

  1. Primary

     1. To determine the effect of QBECO SSI on clinical remission, as measured by abdominal pain and soft-stool frequency, at the end of the maintenance period
     2. To determine the effect of QBECO SSI on endoscopic remission at the end of the maintenance period
     3. To determine the safety and tolerability of QBECO SSI treatment, as measured by safety laboratory assessments, vital signs, frequency and severity of adverse events and physical examinations.
  2. Secondary

     1. To determine the effect of QBECO SSI on clinical remission and endoscopic remission among subjects who were in clinical or endoscopic remission at the end of induction.
     2. To determine the effect of QBECO SSI on abdominal pain score at the end of maintenance period (i.e., change from baseline)
     3. To determine the effect of QBECO SSI on soft-stool score at the end of maintenance period (i.e., change from baseline)To determine the effect of QBECO SSI on endoscopic response at the end of the maintenance period
     4. To determine the effect of QBECO SSI on SES-CD scores at the end of the maintenance period as defined by SES-CD reduction by ≥25% and ≥75% and change from BL
     5. To determine the effect of QBECO SSI on histological activity of CD patients at the end of the maintenance period as defined by 25%, 50% and 75% reduction in global colonic GHAS and RHI
     6. To determine the effect of QBECO SSI on simultaneous clinical and endoscopic remission at the end of the maintenance period

ELIGIBILITY:
Inclusion Criteria:

* Participants who have an established diagnosis of ileal, ileocolonic or colonic CD of at least 3 months duration prior to planned initial dose as determined by endoscopic imaging.
* Participants with a recorded Simple Endoscopic Score for Crohn's Disease (SES-CD) score ≥7 at screening. Subjects with ileitis only will require SES-CD score ≥4.
* Participants with:

  1. a minimum total abdominal pain score above 21 for 7 consecutive days during the screening period, as rated on an 11-point numeric rating scale, OR
  2. a minimum total number of liquid/very soft stools above 10, (Type 6 or 7 as rated by the BSFS), for 7 consecutive days during the screening period.
* Participants may be receiving a therapeutic dose of the following medications:

  1. Oral 5-ASA compounds provided that the dose has been stable for the 2 weeks immediately before screening visit.
  2. Oral corticosteroid therapy (prednisone at a stable dose ≤ 30 mg/day, budesonide at a stable dose ≤ 9 mg/day, or equivalent steroid) provided that the dose has been stable for the 2 weeks before screening visit.
  3. Probiotics provided that the dose has been stable for the 2 weeks immediately before screening visit.
  4. Anti-diarrheal medications (e.g., loperamide, diphenoxylate with atropine) for control of chronic diarrhoea.
  5. Azathioprine or 6-MP provided that the dose has been stable for the 8 weeks immediately before screening visit.
  6. Methotrexate provided that the dose has been stable for the 8 weeks immediately before screening visit.
  7. Antibiotics used for the treatment of CD (i.e., ciprofloxacin, metronidazole) provided that the dose has been stable for at least 2 weeks before screening visit.
* All men must agree to use contraception during the treatment period and for at least 2 months after the last dose of study medication and refrain from donating sperm during this period.
* Women will be eligible to participate if they are not pregnant , not breastfeeding, and at least one of the following conditions applies:

  i. Not a woman of childbearing potential (WOCBP) OR ii. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 2 months after the last dose of study medication.
* Capable of giving signed informed consent as described in Section 11.1.3 - Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Consent to genetic sample collection is not mandatory for inclusion.

Exclusion Criteria:

1. Medical Conditions

   * Evidence of abdominal abscess during screening.
   * Extensive colonic resection or subtotal or total colectomy.
   * Diagnosis of short bowel syndrome.
   * Have received tube feeding, defined formula diets, or parenteral alimentation within 21 days before screening visit.
   * Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
   * Evidence of or treatment for C. difficile infection or other intestinal pathogen within 28 days before screening visit.
   * Currently require or are anticipated to require major surgical intervention for CD (e.g., bowel resection) during the first 26 weeks of the study.
   * History or evidence of adenomatous colonic polyps that have not been removed.
   * Chronic hepatitis B or C infection.
   * Any identified congenital or acquired immunodeficiency (e.g., common variable immunodeficiency, human immunodeficiency virus infection, organ transplantation).
   * Any live vaccinations within 30 days before screening visit except for the influenza vaccine.
   * Women who are lactating or have a positive urine pregnancy test during the Screening period.
   * Any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, GI, genitourinary, haematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the Investigator, would confound the study results or compromise subject safety.
   * Any surgical procedure requiring general (e.g., endotracheal) anaesthesia within 30 days before screening visit or is planning to undergo major surgery during the first 26 weeks of the study.
   * A current or recent colorectal histopathology report that shows positive dysplasia within the past 3 years from final screening visit.
   * Any history of malignancy, except for the following: (a) adequately-treated non-metastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year before screening visit; and (c) history of cervical carcinoma that has been adequately treated and that has not recurred for at least 3 years before screening visit. Subjects with remote history of malignancy (e.g., > 5 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with Qu Biologics' sponsor on a case-by-case basis before enrolment.
2. Prior Concomitant therapy

   * Within 30 days before screening visit, have received any of the following for the treatment of underlying disease:

     1. Non-biologic therapies (e.g., cyclosporine, thalidomide) other than those specifically listed above
     2. A non-biologic investigational therapy
     3. An approved non-biologic therapy in an investigational protocol
   * Within 60 days before screening visit, have received any of the following:

     1. Infliximab
     2. Adalimumab
     3. Certolizumab pegol
     4. Any other investigational or approved biological agent, other than local administration for non-IBD conditions (e.g., intra-ocular injections)
   * Use of topical (rectal) treatment with 5-ASA or corticosteroid enema/suppositories within 2 weeks before screening visit.
3. Diagnostic assessments

   - Any of the following laboratory abnormalities during the Screening period:
   1. Haemoglobin level < 9 g/dL (90 g/L)
   2. White blood cell (WBC) count < 3 x 103/µL (3 x 109/L)
   3. Lymphocyte count < 0.5 x 103/µL (0.5 x 109/L)
   4. Platelet count < 100 x 103/µL (100 x 109/L) or > 1200 x 103/µL (1200 x 109/L)
   5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x the upper limit of normal (ULN)
   6. Alkaline Phosphatase > 3 x ULN
   7. Serum creatinine > 2 x ULN
   8. Albumin < 2.0 g/dL (< 20 g/L)
4. Prior/Concurrent Clinical Study Experience

   - Previous exposure to QBECO SSI or any other Qu Biologics' SSI.
5. Other Exclusions

   * Known or suspected hypersensitivity to any component of the study treatment (i.e., killed whole cell bacterial vaccines).
   * Daily use of narcotic drugs containing opiates (such as morphine, codeine, etc.) for pain control.
   * A current or recent diagnosis (within the past 12 months) of alcohol dependence or illicit drug use, with the exception of medicinal marijuana prescribed by a physician.
   * Active psychiatric problems that, in the Investigator's opinion, may interfere with compliance with the study procedures.
   * Unable to attend all the study visits or comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Lead-In: Selection of Induction Point | week 26
  To determine whether Week 26 provides superior endoscopic healing outcomes compared to Week 16
Main: Clinical Remission at Induction | week 16 or 26
  To determine the effect of QBECO SSI on clinical remission, as measured by abdominal pain and soft-stool frequency, at the end of the induction period
Main: Endoscopic Remission (SES-CD score of 0-2) at Induction | week 16 or 26
  To determine the effect of QBECO SSI on endoscopic remission at the end of the induction period
Main: Clinical Remission | week 52
  To determine the effect of QBECO SSI on clinical remission, as measured by abdominal pain and soft-stool frequency, at the end of the maintenance period
Main: Endoscopic Remission (SES-CD score of 0-2) | week 52
  To determine the effect of QBECO SSI on endoscopic remission at the end of the maintenance period
Incidence of Adverse events (Safety Evaluation) | week 56
  To evaluate the incidence of adverse events (safety and tolerability) as measured by frequency and severity of adverse events.

SECONDARY OUTCOMES:
Lead-in: Endoscopic remission (SES-CD score of 0-2) | week 52
  To determine the effect of QBECO SSI on endoscopic remission at the end of 52 weeks of treatment
Main: Endoscopic Remission (SES-CD score of 0-2) Subpopulation | week 52
  To determine the effect of QBECO SSI on endoscopic remission among subjects who were in clinical or endoscopic remission at the end of induction.
Main: Clinical Remission Subpopulation | week 52
  To determine the effect of QBECO SSI on clinical remission among subjects who were in clinical or endoscopic remission at the end of induction.
Main: Abdominal Pain (11-point numerical rating scale (from 0 (no pain) to 10 (maximum pain))) | week 52
  To determine the effect of QBECO SSI on abdominal pain score at the end of maintenance period (i.e., change from baseline)
Main: Soft-stool Score | week 52
  To determine the effect of QBECO SSI on soft-stool score at the end of maintenance period (i.e., change from baseline)
Main: Abdominal Pain (11-point numerical rating scale (from 0 (no pain) to 10 (maximum pain))) at Induction | week 16 or 26
  To determine the effect of QBECO SSI on abdominal pain score at the end of the induction period (i.e., change from baseline)
Main: Soft-stool score at Induction | week 16 or 26
  To determine the effect of QBECO SSI on soft-stool score at the end of the induction period (i.e., change from baseline)
Main: SES-CD Scores | week 52
  To determine the effect of QBECO SSI on SES-CD scores at the end of the maintenance period as defined by SES-CD reduction by ≥25% and ≥75% and change from baseline
Main: Histological Activity | week 52
  To determine the effect of QBECO SSI on histological activity of CD patients at the end of the maintenance period as defined by 25%, 50% and 75% reduction in global colonic Global Histologic Disease Activity Score (GHAS) and Robarts Histological Index (RHI)
Main: SES-CD Scores at Induction | week 16 or 26
  To determine the effect of QBECO SSI on SES-CD scores at the end of the induction period as defined by SES-CD reduction by ≥25% and ≥75% and change from baseline
Main: Histological Activity at Induction | week 16 or 26
  To determine the effect of QBECO SSI on histological activity of CD patients at the end of the induction period as defined by 25%, 50% and 75% reduction in global colonic Global Histologic Disease Activity Score (GHAS) and Robarts Histological Index (RHI)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Fraser Clinical Trials, New Westminster, British Columbia
  - G.I. Research Institute, Vancouver, British Columbia
  - McMaster University Medical Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No